CLINICAL TRIAL: NCT01196663
Title: Clinical Evaluation of TMS (Temperature Monitoring System) Performance
Brief Title: Comparison of the Performance of TMS-thermometer With Standard Esophageal or Urine Bladder Thermometer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Avi Weissman MD, Rambam Health Care Campus
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TMS-thermometer-CTIL
Record Dates: First submitted 2010-07-28; First posted 2010-09-08 (Estimated); Last update posted 2010-09-22 (Estimated); Status verified 2010-07

CONDITIONS: to Evaluate the Performance of the TMS Thermometer and; Improve Its Algorithm
Keywords: TMS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Intraoperative temperature measurement by TMS thermometer — Measurements will be taken from the patient's body using a biocompatible patch that will transfer data to the receiving unit. The patch will be sterilized before each surgery.
Device: Esophageal or urinary bladder temperature measurement — Standard temperature measurement as is being measured from patients during surgery today

SUMMARY:
This Clinical study is preformed in order to estimate the performance of the TMS thermometer and to make a final tuning of the thermometer mathematical algorithm.

Body temperature of men, women and children will be measured using the TMS thermometer.

Each Patient will be measured both with the TMS thermometer and with an esophageal or urinal thermometer as a reference.

DETAILED DESCRIPTION:
Temperature measurement is vital during surgery. Accurate temperature reading can indicate patient's condition and alarm if something is wrong.

Nowadays, during surgeries temperature is measured mostly using an esophageal or a urinal thermometer, both of which are invasive, therefore they complicate the procedure and require time and activity of the medical stuff.

The TMS thermometer combines a noninvasive, biocompatible patch, which is attached to the body, and a receiving unit, which is placed near the body or the vital signs monitors and receives data from the patch. There is no connection between the body and the receiving unit. The measurement is based on a conductive sensor that measures the skin temperature and applies special algorithm in order to calculate the core body temperature.

The purpose of this clinical study is to evaluate the performance of the TMS thermometer and improve its algorithm by comparing its measurement to the esophageal or urinal temperature measurement

ELIGIBILITY:
Inclusion Criteria:

* Men, women and children that are about to have surgery which requires temperature monitoring.
* An informed consent was signed by the patient or his guardian.

Exclusion Criteria:

* The medical staff decides that the patient can't participate.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between TMS and the esophageal/urinary temperature measurements | The results of this study will be presented in 6 months from today (an average)
  TMS will track patient's temperature during the operation concurrently with esophageal and/or urinary temperature sensor. Correlation will be calculated between both temperature measurement methods and tracking ability of the changes in patient's temperature during the operation will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Avi Weissman, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Dept of anesthesiology -Rambam health care campus, Haifa, Israel